CLINICAL TRIAL: NCT04183231
Title: Pharmacokinetics of Advantage Anti-Caries Varnish
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advantage Silver Dental Arrest, LLC (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-04-05
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-07

CONDITIONS: Dental Caries
Keywords: adults; povidone iodine; sodium fluoride
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Open label exposure--response study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-caries varnish (Experimental): topical dental varnish, 10% PVP-I, 2.5% NaF, topical application to teeth, 0.4 ml, single application
  Interventions: Drug: Anti-caries varnish

INTERVENTIONS:
Drug: Anti-caries varnish — topical tooth varnish

SUMMARY:
The study aim is to characterize the kinetics of iodine and fluoride following topical application of a combined PVP-I and NaF anti-dental caries varnish in healthy adults.

DETAILED DESCRIPTION:
The study was to characterize serum iodine and fluoride levels over 24 hours after application of a topical dental varnish in healthy adults 23 to 57 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18 y and older, at least 20 teeth, not taking prescription or OTC medications.

Exclusion Criteria:

* Pregnant, weighed less than 110 pounds, had oral mucositis, ulcerative lesions, sensitivity to shellfish or iodine or fluoride varnish, or had known hypothyroidism, hyperthyroidism, dermatitis herpetiformis, hypocomplementemic vasculitis, nodular thread with heart disease, multi nodular goiter, Graves disease, or autoimmune thyroiditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lin, PhD, Principal Investigator — University of Washington School of Pharmacy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin YS, Rothen ML, Milgrom P. Pharmacokinetics of Iodine and Fluoride following Application of an Anticaries Varnish in Adults. JDR Clin Trans Res. 2018 Jul;3(3):238-245. doi: 10.1177/2380084418771930. Epub 2018 Apr 25. PMID 30938600

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-caries Varnish
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Observed Iodine Tmax
Description: Time to maximum serum concentration of iodine in hours
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
hours | 1.7 (0.7)

2. Primary Outcome: Observed Iodine Cmax
Description: Maximum serum concentration of iodine in ng/mL
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
ng/mL | 111 (36)

3. Primary Outcome: Observed Iodine Baseline-Corrected Cmax
Description: Maximum serum concentration of iodine in ng/mL
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
ng/mL | 57 (33)

4. Primary Outcome: Observed Iodine Baseline-Corrected AUC
Description: Area under the Curve for observed iodine in ng*h/mL
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng-h/mL
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
ng-h/mL | 539 (315)

5. Primary Outcome: Observed Iodine Total Urinary Recovery
Description: Total urinary recovery in milligrams observed
Time Frame: baseline to 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
mg | 1.26 (0.71)

6. Primary Outcome: Iodine t1/2
Description: Terminal elimination half-life of iodine in hours
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
hours | 5.5 (1.4)

7. Primary Outcome: Observed Fluoride Tmax
Description: Time to maximum serum concentration in hours
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
hours | 0.8 (0.3)

8. Primary Outcome: Observed Fluoride Cmax
Description: Maximum serum concentration of fluoride in ng/mL
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
ng/mL | 76 (36)

9. Primary Outcome: Observed Fluoride Baseline-Corrected Cmax
Description: Maximum serum concentration of iodine in ng/mL
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
ng/mL | 60 (34)

10. Primary Outcome: Observed Fluoride AUC
Description: Area under the Curve for observed fluoride in ng*h/mL
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng-h/mL
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
ng-h/mL | 703 (350)

11. Primary Outcome: Observed Fluoride Baseline-Corrected AUC
Description: Area under the Curve for observed fluoride in ng*h/mL
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng-h/mL
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
ng-h/mL | 315 (206)

12. Primary Outcome: Fluoride t1/2
Description: Terminal elimination half-life in hours for fluoride
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
hours | 3.1 (1.6)

13. Primary Outcome: Observed Fluoride Total Urinary Recovery
Description: Total urinary recovery in milligrams observed
Time Frame: baseline to 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Anti-caries Varnish
Number analyzed (Participants) | 16
mg | 2.51 (1.28)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Anti-caries Varnish
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT04183231/Prot_SAP_000.pdf